CLINICAL TRIAL: NCT05074342
Title: Guiding Primary Care Diabetic Retinopathy Screening in Canada Through the Use of Provincial Healthcare Administrative Data
Brief Title: Project Open - Use of Administrative Health Data to Increase Diabetic Retinopathy Screening
Status: Enrolling by invitation | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: South Riverdale Community Health Centre (Unknown); Flemingdon Health Centre (Unknown); Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, Michael Brent, MD, FRCSC Principal Investigator -Clinical Lead, University Health Network, Toronto
Other Study IDs: 8 Sep 2020
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Diabetic Retinopathy
Keywords: Administrative data; Screening
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early detection through regular diabetic retinopathy screening (DRS) is an effective method of preventing vision loss by enabling earlier intervention and timely treatment. It is recommended that all people with diabetes receive regular DRS, either annually or bi-annually. Current DRS practice in Canada, however, falls remarkably short of recommended DRS rates resulting in preventable vision loss.

In this project the investigators use population health-based approach to diabetes care. Linked provincial administrative data will be leveraged to consistently identify all those that have not had DRS in 425 days with the goal to improve outcomes, equity and potentially reduce the cost of care delivery.

DETAILED DESCRIPTION:
Diabetic Retinopathy (DR) is the leading cause of blindness in working age Canadians. Canada fall remarkably short of this recommended rate resulting in many Canadians with preventable vision loss, despite the availability of ophthalmology and/or optometry services covered by provincial health insurance plans. It is estimated that in Ontario alone that up to 40% of individuals with diabetes have not had their eyes screened for retinopathy. To address the low rate, tele-ophthalmology or Tele-Retina, using telemedicine resources, has been an approach used in a variety of primary health care settings in urban, rural and remote areas across Canada. In the United Kingdom, a population-based approach to this issue have been taken and have lowered the unscreened rate, resulting in diabetic retinopathy no longer being the leading cause of blindness in working age individuals. New strategies are required to identify, engage, and provide ongoing monitoring to those requiring DR screening in Ontario.

The electronic medical records in doctors' offices do not receive information about the status of patients with diabetes retinopathy screening status. This information only exists through provincial data and public insurance system billings. Using administrative health data, the investigators developed a population-based approach to DR screening at community health centres (CHCs). Patients with diabetes who have not had DR screening in 425 days have been identified using linked provincial and community-based datasets.

Through the linking of the Alliance for Healthier Communities dataset with other Ontario healthcare administrative databases held at Institute for Clinical Evaluative Sciences (IC/ES), the investigators have identified clients within the CHC that have not had eyes checked for signs of retinopathy by an ophthalmologist or optometrist within the previous 425 days. This data is transferred to the CHC and the identified clients will then be called to let them know about the importance of having their eyes examined and to see if they are interested in participating in the study. Through the Diabetes Eye Screening Program, Tele-Retina will be made available through referral. If individuals are not interested in this program, patients will be encouraged to seek alternate ophthalmology or optometry services.

Qualitative semi-structured interviews examining diabetic retinopathy screening and the Tele-Retina process at the CHC, including facilitators and barriers towards diabetes care, specifically eye care, will be conducted. The investigators will be interviewing patients, caregivers, healthcare practitioners, CHC staff, management and policy decision-makers.

The intervention of providing provincial-level diabetic retinopathy status to primary health care settings will be evaluated using a mixed-methods implementation-effectiveness hybrid approach. Evaluation will be conducted concurrently with the study intervention to evaluate its effectiveness, cost-effectiveness, implementation barriers and key success factors. The evaluation will consist of 4 main components of 1) an implementation study, 2) a policy study, 3) clinical evaluation and 4) economic evaluation studies.

Our overall objectives for the study are to:

1. Increase the number of screened individuals who are at risk for DR within the primary care settings, and to refer to treatment those at risk of vision loss;
2. Evaluate implementation and policy barriers associated with the transfer and use of healthcare administrative data related to DR, at a primary care level and DR screening in general;
3. Evaluate patient and provider experience and attitudes with the initiative, including sex and gender and socioeconomic factors;
4. Describe the severity of diabetic retinopathy in those individuals who agree to be screened;
5. Examine the healthcare resource utilization and costs and cost-effectiveness associated with the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Type 1 or type 2 diabetes as determined through linked provincial healthcare administrative datasets or primary care data using algorithms similar to provincial methods.
3. Attended the primary health care setting, with at least 1 visit to the centre within the past 10 years

Exclusion Criteria:

1. Individuals identified as having received DRS (in the previous 425 days) by an ophthalmologist and/or optometrist or tele-ophthalmology/Tele-Retina.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with type 1 or type 2 diabetes, who have attended a primary healthcare setting at CHCs, and through the use of provincial administrative data is identified as the patient who has not had their eyes screened within the past 425 days.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The provision of a DRS status list to primary health care settings will increase the rate of annual DR screening in patients with type 1 or type 2 diabetes who have attended the centres. | 425 days
  To increase the screening rate of individuals who are at risk for DR within the primary care settings, and to refer to treatment those at risk of vision loss.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontarioa, Canada